CLINICAL TRIAL: NCT06812377
Title: Comparative Study Between Different Mobilization Techniques for Patients With Chronic Tennis Elbow
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammad Moustafa Aldosoukki Hegazy, dr, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCBR-393/2024; 2024/03/31970 (Other Grant/Funding Number: Prince Sattam bin Abdulaziz University)
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Tennis Elbow
Keywords: Tennis elbow, Grip strength, Pain pressure threshold , Nerve mobilization , Maitland mobilization, Mulligan mobilization
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): maitland mobilization Posteroanterior mobilization of the radial head in motion. This method is gliding over the radial head posteriorly to anteriorly while the patient executes (and relaxes) the painful action (e.g., clutching). Repeat the method six to ten times if there is a noticeable increase in your ability to grip without pain
  Interventions: Other: Maitland joint mbilization
- Group (B) (Active Comparator): mulligan mobilization Using this approach, the patient performs (and relaxes) the painful action (e.g., clutching) while a lateral humeroulnar auxiliary glide is applied and maintained. If you notice a noticeable increase in your ability to grip without pain, repeat the method six to ten times. You can use a belt to help you glide.Three sets of it were performed, with a 30-second break in between [44].
  Interventions: Other: mulligan mobilization
- Group (c) (Experimental): radial nerve mobilization
  Interventions: Other: radial nerve mobilization

INTERVENTIONS:
Other: Maitland joint mbilization — Posteroanterior mobilization of the radial head in motion. This method is gliding over the radial head posteriorly to anteriorly while the patient executes (and relaxes) the painful action (e.g., clutching). Repeat the method six to ten times if there is a noticeable increase in your ability to grip without pain
  Arms: group A
Other: mulligan mobilization — Using this approach, the patient performs (and relaxes) the painful action (e.g., clutching) while a lateral humeroulnar auxiliary glide is applied and maintained. If you notice a noticeable increase in your ability to grip without pain, repeat the method six to ten times. You can use a belt to help you glide.Three sets of it were performed, with a 30-second break in between
  Arms: Group (B)
Other: radial nerve mobilization — The subjects will be placed in a reclining supine position. The arm will be internally rotated, the wrist, thumb, and fingers will be flexed, the shoulder girdle will be depressed, and the elbow will be stretched. Elbow flexion and wrist extension will be used to maintain shoulder depression after the radial nerve will be strained by these motions. Before beginning the gentle elbow extension test, the subject's wrist and fingers will be stabilized. The elbow will be then gently extended for about two seconds, just into the range where the participant felt tension but no pain, and then flexed. In a single session, three sets of six to eight oscillations will be executed
  Arms: Group (c)

SUMMARY:
Background: Tennis elbow is a common musculoskeletal disorder affecting the functional activities of daily living through common extensor tendinopathy. There is a limited knowledge about neural restriction as a source of movement limitation in patients with tennis other than enriched joint mobilization techniques knowledge.

Objectives: This study will be designed to determine the efficacy of adding different mobilization techniques along with eccentric exercises on elbow pain intensity, functional disability, hand grip strength and pain pressure in patients with chronic tennis elbow.

Methods: Forty five patients with lateral epicondylitis with their ages ranged from 18 and 45 more than six weeks will be randomly assigned into three groups. Group A will receive Maitland joint mobilization techniques. Patients in group B will receive Mulligan mobilization techniques while patient in group C will receive radial nerve mobilization.. Both groups will receive eccentric exercises for wrist extensors . Patients will be treated three session per week for four week and they will be evaluated pre and post treatment for pain severity using by visual analogue scale, level of functionality by DASH questionnaire, hand grip strength by hand held dynamometer and pressure pain threshold(PPT) by pressure algometer.

Results: All the outcome variables will be assessed at baseline and 4weeks following the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* This study will include individuals between the ages of 18 and 45 who have been diagnosed with lateral epicondylitis based on positive results from the Mill's and Cozen's tests. The participants must also have complaints of local tenderness at the elbow that lasts longer than six weeks. Additionally, to complete the assessment and get treatment, the participants' elbow must have a full extension range of motion

Exclusion Criteria:

* Individuals diagnosed with cervical radiculopathy, upper thoracic outlet syndrome, rheumatoid arthritis, myositis ossificans, carpal tunnel syndrome, recent upper limb trauma, elbow immobilization, steroid injection administration within the previous six months, and any history of physical therapy administered within the previous six months were excluded from the study. Furthermore, participation will not be permitted for anyone who has previously experienced discomfort because of their profession

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
elbow pain | At baseline and after 4 weeks
  Assessment of pain intensity will be measured by visual analogue scale (VAS) which consists of a vertical line (0-10) where one end refers to no pain while the other end refers to great pain.) It is a reliable test for literate and illiterate patients 0.94I,0.71 respectively)
Hand grip strength | At baseline and after 4 weeks
  To assess hand grip strength, In order to assess grip strength painlessly, the patient will comfortably sit with their arm at their side, their shoulder adducted and neutrally rotated, their elbow flexed to 90 degrees [38], their forearm in a neutral position, their wrist between 0 and 30 degrees of extension, and their ulnar deviation between 0 and 15 degrees. The greatest grip contraction, expressed in kilograms, shall be noted when no discomfort is felt. The patient will squeeze for three to five seconds, as hard as they can. Multiple trials will be conducted, with an average of three repetitions recorded and a gap of approximately 15 seconds between each trial, to mitigate the possible effect of muscle fatigue

SECONDARY OUTCOMES:
pain pressure threshold | At baseline and after 4 weeks
  Pain Pressure Threshold (PPT) will be measured by pressure algometer by applying the probe tip on the most sensitive poin. Also, three trials will be given, and the average will be taken [39].
  A portable device called a pressure algometer is used to measure the pressure-pain threshold. The lowest pressure value at which a person feels pain is known as the pressure-pain threshold [40]. One accurate way to gauge someone's level of discomfort is by using their pressure-pain threshold [41]. A force gauge with a spring-operated plunger is called an algometer. The gauge is fastened to a short metal pole with a rubber tip that is circular and has a diameter of 1 cm. The unit of calibration for the instrument is kilograms of pressure per square centimeter (kg/cm2). The gauge measures between 0 and 10 kg/cm^2. The gadget can be reset to 0 to take a new measurement once one has been taken
functionality | At baseline and after 4 weeks
  Assessment of level of functionality:
  A 30-item disability/symptom scale that evaluates the patient's health during the preceding week is the main component of the DASH [36]. The questions include how difficult it is to perform different physical activities due to an arm, shoulder, or hand problem (21 items), how severe each pain symptom is, how much pain, tingling, weakness, or stiffness is related to a particular activity (5 items), and how the problem affects social activities, work, sleep, and one's self-image (4 items). For every item, there are five possible responses. A scale score ranging from 0 (no impairment) to 100 (full disability) (most severe disability) is then obtained by adding the scores for each component

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vicenzino B, Paungmali A, Teys P. Mulligan's mobilization-with-movement, positional faults and pain relief: current concepts from a critical review of literature. Man Ther. 2007 May;12(2):98-108. doi: 10.1016/j.math.2006.07.012. Epub 2006 Sep 7. PMID 16959529
- [Background] Coombes BK, Bisset L, Vicenzino B. Management of Lateral Elbow Tendinopathy: One Size Does Not Fit All. J Orthop Sports Phys Ther. 2015 Nov;45(11):938-49. doi: 10.2519/jospt.2015.5841. Epub 2015 Sep 17. PMID 26381484
- [Background] Dorf ER, Chhabra AB, Golish SR, McGinty JL, Pannunzio ME. Effect of elbow position on grip strength in the evaluation of lateral epicondylitis. J Hand Surg Am. 2007 Jul-Aug;32(6):882-6. doi: 10.1016/j.jhsa.2007.04.010. PMID 17606071